CLINICAL TRIAL: NCT03443830
Title: Phase 1 First in Human, Time Lagged, Parallel-Group, Single Ascending Dose Study of Tyzivumab in Healthy Adult Volunteers
Brief Title: Safety and Tolerability of an Antibody Against Zika Virus (Tyzivumab) in Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tychan Pte Ltd. (Industry)
Collaborators: Duke-NUS Graduate Medical School (Other); Singapore Clinical Research Institute (Other); National University of Singapore (Other); National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZKT-001
Record Dates: First submitted 2018-02-08; First posted 2018-02-23 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Treatment of Acute Zika Virus Infection
Keywords: Zika virus; Tyzivumab; Monoclonal antibody; Infectious diseases; Phase 1A first in human study; Singapore
MeSH Terms: conditions — Zika Virus Infection; Communicable Diseases

STUDY DESIGN:
Intervention Model Description: Time Lagged, Parallel-Group, Single Ascending Dose Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- 0.2 mg/kg (Experimental): Subject will be administered with 0.2 mg/kg of Tyzivumab via IV infusion over a period of 30 minutes.
  Interventions: Drug: Tyzivumab
- 0.5 mg/kg (Experimental): Subject will be administered with 0.5 mg/kg of Tyzivumab via IV infusion over a period of 30 minutes.
  Interventions: Drug: Tyzivumab
- 1 mg/kg (Experimental): Subject will be administered with 1 mg/kg of Tyzivumab via IV infusion over a period of 30 minutes.
  Interventions: Drug: Tyzivumab
- 5 mg/kg (Experimental): Subject will be administered with 5 mg/kg of Tyzivumab via IV infusion over a period of 30 minutes.
  Interventions: Drug: Tyzivumab
- 10 mg/kg (Experimental): Subject will be administered with 10 mg/kg of Tyzivumab via IV infusion over a period of 30 minutes.
  Interventions: Drug: Tyzivumab
- 20 mg/kg (Experimental): Subject will be administered with 20 mg/kg of Tyzivumab via IV infusion over a period of 30 minutes.
  Interventions: Drug: Tyzivumab

INTERVENTIONS:
Drug: Tyzivumab — Tyzivumab Injection, (100 mg/5 mL/Vial), Zika Virus (ZIKV) Monoclonal Antibody (mAb) Infused over 30 minutes
  Other Names: TY008

SUMMARY:
Zika virus (ZIKV) infection is a new emerging arbovirus disease, caused by the same vector that transmits Dengue virus, Aedes aegypti. ZIKV is a growing public health problem, rapidly spreading throughout the continents since the first epidemic was reported in the French Polynesian islands.

Currently, there are several ZIKV vaccine candidates in clinical trials. However, no ZIKV therapy (biologic or small molecule) has advanced to clinical trials. Tyzivumab will be the first therapeutic in the world, specifically targeting ZIKV, to enter clinical trials.

This is a Phase 1, first in human, time-lagged, parallel-group, single dose ascending (6 dose cohorts), Tyzivumab, ZIKV monoclonal antibody (mAb), study to be conducted in 24 flaviviral naïve healthy adult volunteers.

Tyzivumab will be administered once through single IV infusion over 30 minutes. Total duration of study participation is estimated at approximately 98 days from the date of screening. Post-trial monitoring through weekly telephone calls will continue from Day 85 post-dose onwards for another three (3) more months.

The main objective of this study is to evaluate safety of Tyzivumab in healthy adult volunteers through assessment of subject vital signs, clinical laboratory results, ECG, presence/absence of AE/SAE, PK and ADA.

DETAILED DESCRIPTION:
Dose escalation in this study will include 24 healthy volunteers in six (6) dose cohorts:

* 0.2 mg/kg, N = 2
* 0.5 mg/kg, N = 2
* 1 mg/kg, N = 2
* 5 mg/kg, N = 6
* 10 mg/kg, N = 6
* 20 mg/kg, N = 6

A minimum of 20-hour interval from the first dosing must take place before the second subject can be dosed within each cohort. No such time interval will be required for dosing of subsequent subjects (third subject onwards) within the same cohort.

Dose escalations will be guided by review of clinical signs, adverse events (AEs), and laboratory tests of the prior group (up to Day 7 after dosing) by a safety monitoring committee.

In order to assess the safety and tolerability of an intravenous (IV) infusion of Tyzivumab when given to healthy adult volunteers, the following vital signs and tests will be performed:

* Blood Pressure
* Pulse Rate
* Respiratory Rate
* Body Temperature
* ECG
* Urinalysis
* Serum Chemistry
* Haematology

In order to assess Tyzivumab pharmacokinetics (only for doses 1 mg/kg, 5 mg/kg, 10 mg/kg & 20 mg/kg), the following parameters will be measured:

* maximum concentration (Cmax)
* time to maximum concentration (Tmax)
* area under the curve extrapolated to infinity (AUC0-∞)
* AUC calculated from time of administration to the last measurable concentration (AUC0-last)
* half-life (t1/2)
* volume of distribution (Vd)
* clearance [CL] in serum PK will be assessed at pre-dose, 0.5 h, 1 h, 2 h, 4 h, 8 h, 24 h, 48 h, 72 h, 120 h, Day 7, Day 14, Day 28, Day 56 and Day 84.

The presence and extent of anti-drug antibody (ADA) production in response to dosing with Tyzivumab will also be assessed at pre-dose, Day 14, Day 56 and Day 84.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet all the following criteria to be enrolled:

1. Adult healthy volunteers, aged 21 to 45, men or women

   a. Women must fulfil one (1) of the following criteria: i. Post-menopausal; either amenorrhea ≥ 12 months or follicle stimulating hormone > 40 mIU/mL ii. Surgically sterile; hysterectomy, bilateral oophorectomy, or tubal ligation iii.Women of childbearing potential participating in heterosexual sexual relations must be willing to use adequate contraception from screening day until 100 days post-infusion b. Male subjects who are non-vasectomized (or vasectomized less than six (6) months prior to dosing) and have female partners of childbearing potential must be willing to use an effective birth control method when having heterosexual intercourse, from screening day until 100 days post-infusion
2. Subjects negative for antibodies to flaviviruses as measured by a commercially available Dengue virus IgG enzyme-linked immunosorbent assay (ELISA) diagnostic kit
3. Subjects negative for human immunodeficiency virus (HIV), Hepatitis B virus (HBV) and Hepatitis C virus (HCV)
4. Subjects who are willing to comply with the requirements of the study protocol and attend scheduled visit
5. Subjects who give written informed consent approved by the Ethical Review Board governing the site
6. Satisfactory baseline medical assessment as assessed by physical examination and normal laboratory values or minor variations that are acceptable for study entry
7. Accessible vein in the forearm for blood collection

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

1. History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, neuropsychiatric, or immunosuppressive disorders
2. Evidence of clinically significant anaemia (HB < 10 g/dL) or any other significant active haematological disease, or having donated > 450 mL of blood within the past three (3) months
3. Evidence of substance abuse, or previous substance abuse
4. Participation or planned participation in a study involving the administration of an investigational compound within the past four (4) months or during this study period
5. Planned administration of any vaccine not foreseen by the study protocol 12 weeks before first dosing day and up to four (4) months after dosing
6. Receipt of immunoglobulins and/or any blood products within nine (9) months of study enrolment or planned administration of any of these products during the study period
7. History of any reaction to monoclonal antibodies
8. Pregnant or lactating women, or women of childbearing potential who are unwilling to use adequate contraception
9. Any condition that, in the opinion of the investigator, would complicate or compromise the study or well-being of the subject

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2018-12-04 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Event (Safety and Tolerability) | 84 days
  Presence or absence of infusion reaction (hypersensitivity / anaphylaxis / etc.) in dose cohorts.

SECONDARY OUTCOMES:
Maximum Concentration (Cmax) - Pharmacokinetic Assessment | Pre-dose, 0.5 hour, 1 hour, 2 hour, 4 hour, 8 hour, 24 hour, 48 hour, 72 hour, 120 hour Day 7, Day 14, Day 28, Day 56 and Day 84.
  Constant monitoring of the levels of antibody in subject sera through various time points as stated below would help elucidate the maximum concentration (Cmax) of Tyzivumab in human serum.
Time to Maximum Concentration (Tmax) - Pharmacokinetic Assessment | Pre-dose, 0.5 hour, 1 hour, 2 hour, 4 hour, 8 hour, 24 hour, 48 hour, 72 hour, 120 hour Day 7, Day 14, Day 28, Day 56 and Day 84.
  Constant monitoring of the levels of antibody in subject sera through various time points as stated below would help elucidate the time to maximum concentration (Tmax) of Tyzivumab in human serum.
Area Under the Curve Extrapolated to Infinity (AUC0-∞) - Pharmacokinetic Assessment | Pre-dose, 0.5 hour, 1 hour, 2 hour, 4 hour, 8 hour, 24 hour, 48 hour, 72 hour, 120 hour Day 7, Day 14, Day 28, Day 56 and Day 84.
  Constant monitoring of the levels of antibody in subject sera through various time points as stated below would help elucidate the area under the curve extrapolated to infinity (AUC0-∞) of Tyzivumab.
AUC calculated from time of administration to the last measurable concentration (AUC0-last) - Pharmacokinetic Assessment | Pre-dose, 0.5 hour, 1 hour, 2 hour, 4 hour, 8 hour, 24 hour, 48 hour, 72 hour, 120 hour Day 7, Day 14, Day 28, Day 56 and Day 84.
  Constant monitoring of the levels of antibody in subject sera through various time points as stated below would help elucidate the AUC calculated from time of administration to the last measurable concentration (AUC0-last) of Tyzivumab.
Half-Life (t1/2) - Pharmacokinetic Assessment | Pre-dose, 0.5 hour, 1 hour, 2 hour, 4 hour, 8 hour, 24 hour, 48 hour, 72 hour, 120 hour Day 7, Day 14, Day 28, Day 56 and Day 84.
  Constant monitoring of the levels of antibody in subject sera through various time points as stated below would help elucidate the half-life (t1/2) of Tyzivumab in human serum.
Volume of Distribution (Vd) - Pharmacokinetic Assessment | Pre-dose, 0.5 hour, 1 hour, 2 hour, 4 hour, 8 hour, 24 hour, 48 hour, 72 hour, 120 hour Day 7, Day 14, Day 28, Day 56 and Day 84.
  Constant monitoring of the levels of antibody in subject sera through various time points as stated below would help elucidate the volume of distribution (Vd) of Tyzivumab in human serum.
Clearance [CL] - Pharmacokinetic Assessment | Pre-dose, 0.5 hour, 1 hour, 2 hour, 4 hour, 8 hour, 24 hour, 48 hour, 72 hour, 120 hour Day 7, Day 14, Day 28, Day 56 and Day 84.
  Constant monitoring of the levels of antibody in subject sera through various time points as stated below would help elucidate clearance [CL] of Tyzivumab in human serum.
Anti-Drug Antibody Assessment | Pre-dose, Day 14, Day 56 and Day 84
  To assess the presence or absence of anti-drug antibody (ADA) production in response to dosing with Tyzivumab

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Low, MBBS, Principal Investigator — SingHealth Investigational Medicine Unit
Locations (1):
- SingHealth Investigational Medicine Unit, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided